CLINICAL TRIAL: NCT06886217
Title: Extending the Reach of Evidence-based Practices to Support Student's Attention and Behavior Through Technology
Acronym: CLS-D
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2024-0192; R324A240184 (Other: National Center for Special Education Research, Institute for Education Science)
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Control Condition; Intervention Condition
Keywords: ADHD; school mental health; digital health interventions; implementation science; web-based applications
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Business As Usual (No Intervention): Students in the control condition will receive the usual services their schools provide to students with or at risk for ADHD in grades 2-5.
- Collaborative Life Skills (Experimental): Student, parents, and teachers in the intervention condition will receive the digitally adapted Collaborative Life Skills program.
  Interventions: Behavioral: Collaborative Life Skills dHealth tool (CLS-D)

INTERVENTIONS:
Behavioral: Collaborative Life Skills dHealth tool (CLS-D) — The purpose of this adapted intervention is to integrate digital health (dHealth) technology into the Collaborative Life Skills Program (CLS), an established, school-based behavioral intervention for students with ADHD, to make the program accessible to schools that serve students from low-socioeconomic (SES) backgrounds. Existing evidence-based interventions for students with ADHD are often inaccessible in schools with limited resources to support implementation. By adapting CLS to include a dHealth tool-CLS-D-researchers aim to improve the feasibility of intervention implementation in schools with limited resources and mitigate disparities in access to evidence-based interventions among students with ADHD who are from low-SES backgrounds.
  Other Names: Collaborative Life Skills (CLS) program
  Arms: Collaborative Life Skills

SUMMARY:
The purpose of this study is to integrate digital health (dHealth) technology into the Collaborative Life Skills Program (CLS), an established, school-based behavioral intervention for students with ADHD, to make the program accessible to schools that serve students from low-socioeconomic (SES) backgrounds. Existing evidence-based interventions for students with ADHD are often inaccessible in schools with limited resources to support implementation. By adapting CLS to include a dHealth tool-CLS-D-investigators aim to improve the feasibility of intervention implementation in schools with limited resources and mitigate disparities in access to evidence-based interventions among students with ADHD who are from low-SES backgrounds.

DETAILED DESCRIPTION:
Setting: The research will take place in urban elementary schools in California that receive Title 1 funds to support students who qualify for free or reduced lunch.

Sample: Participants will be SMHPs (one per school) who work half or full time in a school with limited resources that serve students from predominantly low-SES backgrounds, students in grades 2-5 who have ADHD-related impairments (referred to as with or at risk for ADHD), and their parents. In the discovery and design phase, 8 SMHPs, 12 teachers, 12 students, and 12 parents will participate. In the test and refine phase, 4 SMHPs, 24 students, and their parents and teachers, will participate. In the evaluation phase, 12 SMHPs and 72 students and their parents and teachers will participate.

Intervention: The CLS-D intervention, which will be designed to maximize usability, feasibility, and acceptability in schools with limited resources, will include CLS's three evidence-based behavioral treatments for ADHD: behavioral parent training, daily report card with teacher consultation, and child skills training. CLS-D's dHealth tool will consist of a web-based portal with user interfaces for SMHPs, teachers, parents, and students that will be designed to mitigate traditional barriers to accessing services among students with ADHD from low-SES backgrounds. CLS-D will be implemented over a 10-week period and be compatible with various operating systems and devices, including smart phones, tablets, and computers.

Research Design and Methods: During the discovery and design phase, researchers will conduct focus groups with panels of SMHPs, teachers, and students with or at risk for ADHD from low-SES backgrounds and their parents to inform CLS adaptations and dHealth tool development. Researchers and consultants will design an initial prototype of the dHealth tool and adapt CLS-D training, fidelity monitoring, and cost evaluation protocols. During the test and refine phase, researchers will refine the prototype through iterative usability testing with stakeholder panels. Researchers will conduct open trials with SMHPs, students with or at risk for ADHD, and their parents and teachers to test the usability, feasibility, and acceptability of CLS-D, training, fidelity monitoring, and cost evaluation tools. Researchers will also conduct focus groups with participants following the open trials and make final refinements to CLS-D protocols. During the evaluation phase, researchers will use a pilot randomized trial, assigning SMHPs/schools to the CLS-D or control condition, to evaluate the feasibility and promise of CLS-D and the associated costs. The pilot will include two staggered cohorts (fall, spring) in which researchers match pairs of schools based on the proportion of students eligible for free or reduced lunch, the number of students, and racial/ethnic composition. In fall of the school year after the pilot randomized trial, researchers will collect follow-up data on student outcomes.

Control Condition: Students in the control condition will receive the usual services their schools provide to students with or at risk for ADHD in grades 2-5.

Key Measures: Key measures during the discovery and design phase will include a psychometrically validated System Usability Scale (SUS) that SMHPs, teachers, and parents will complete, and a researcher-designed satisfaction scale for SMHPs. During the test and refine phase, key measures will include the SUS, CLS-D usage analytics, and researcher-designed pre/post acceptability and feasibility scales that parents, students, teachers, and SMHPs will complete. During the evaluation and follow-up phase, key measures will include the SUS, acceptability, and feasibility scales; a researcher-developed SMHP fidelity checklist; student-level school records of grades, discipline, and services received; and standardized achievement test scores.

Data Analytic Strategy: For the discovery and design phase, researchers will conduct rapid qualitative content analyses of focus group data using the Rigorous and Accelerated Data Reduction (RADaR) technique and analyze quantitative ratings from the focus groups using descriptive statistics. In the test and refine phase, researchers will use the RADaR technique to analyze qualitative data; use descriptive statistics to analyze process measures, cost measures, and usage analytics; and calculate within-subjects mean differences and Cohen's d effect sizes for pre- and post-assessment data. For the evaluation phase and follow up, researchers will conduct an intent-to-treat analysis using hierarchical linear modeling to examine between-group differences in student outcomes.

Cost Analysis: Researchers will conduct a cost analysis based on a societal perspective using the ingredients approach. Researchers will include information from the cost evaluation tools they will develop during the project, and they will calculate total costs, average cost per student served, the range of costs per student served, and marginal costs per student added once CLS-D is established.

ELIGIBILITY:
Student eligibility criteria:

* Identified by teachers, school mental health professionals, and/or parents with students who have inattention and behavioral problems.
* Must be enrolled in the school districts in the San Diego or San Francisco Bay area
* Must be in 2nd-5th grade
* Placed in a mainstream class
* Eligibility for free or reduced lunch
* Living with a caregiver who is available to participate in treatment
* Must NOT have:

  * Significant visual or hearing impairment
  * Severe language delay, psychosis
  * Pervasive developmental disorder
  * Global intellectual impairment.

Adult participants groups eligibility criteria:

* Parents or caregivers of eligible students can participate in the study.
* School mental health professionals who work with the eligible students can participate in the study.
* Teachers who work with the eligible students can participate in the study.

Exclusion Criteria:

* Researchers will include children with symptoms and impairment of ADHD.
* Researchers would like to involve children in mainstream class placement rather than those who already have services from school (e.g., special education classes).
* Researchers will target those from low SES backgrounds who are eligible for reduced or free lunch.
* All students are expected to be physically healthy, but it should be noted that students with ADHD often have high rates of co-morbid disabilities.
* Furthermore, the researchers would like to invite parents/caregivers, school mental health professionals, and teachers who work with students with ADHD to be involved in focus groups

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | During the 4th week of intervention and following the last week of the 8-week intervention
  This is a psychometrically validated questionnaire will be administered to school mental health professionals, teachers, and parents to assess how easy and user-friendly an interface or digital tool is for its users. This is a 10-item technology agnostic scale assessing technology product usability, with scores above 80 indicating good usability (Brooke, 2014; Lewis & Sauro, 2009, 2018). The SUS has high internal consistency (α=.91) and high convergent validity with a separate rating of usability and user satisfaction (r=.8).
The Feasibility Rating Scale | During the 4th week of intervention and following the last week of the 8-week intervention
  This will be completed by principals, teachers, and school mental health professionals. This measure will contain items regarding the amount of time required to participate in the program, the level of effort needed to identify and enroll students in the program, the availability of physical space needed to run in-person groups, etc. We will query SMHPs weekly (real time) about CLS-D demands on their time, with specific questions regarding their use of the dHealth tool.

SECONDARY OUTCOMES:
Collaborative Life Skills (CLS) intervention fidelity checklist for school mental health providers | Weekly during intervention
  Researchers will rate the school mental health professional's fidelity to the Collaborative Life Skills intervention based on the level of intervention content covered (coverage of each item is rated on a scaled from 0 to 2 where 0 = not covered, 1= partially covered, 2= mostly covered. The quality of intervention implementation regarding school mental health provider's use of clinical skills (e.g., reviewed homework, effectively reviewed handouts, used strategies to promote engagement, asked questions, followed time management guidelines) during each session is also rated on a 1 to 5 scale.

OTHER OUTCOMES:
Student Academics | Baseline; Post-intervention; Follow-up at the end of the first quarter during the subsequent school year
  Students academic and behavioral records will be collected from the school for each student participating in the evaluation phase. These school records include students' grades reports, standardized achievement test scores across academic years enrolled at the school, discipline records across academic years enrolled at the school, and specialized services received across academic years enrolled at the school.
Student Behavioral Progress | Weekly during intervention
  The proportion of school days the school and home Daily Behavioral Report Cards (DBRCs) were implemented each week will be calculated based on the number of completed DBRCs, divided by the overall count of possible days during the week, as we have done in previous trials. School holidays (coded from the online student calendar for each school), child absence, special school events/field trips and substitute teacher days (when noted on the DBRC) will not be included in the overall count of possible school days during the week.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villodas, PhD, Principal Investigator — Department of Psychology, College of Sciences, San Diego State University; Linda Pfiffner, PhD, Principal Investigator — Department of Psychiatry, School of Medicine, University of California San Francisco
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Collaborative Life Skills Digital Mental Health Project (CLS-D) — https://hcfd.sdsu.edu/?page_id=3051
- See also: IES funded research grant: Extending the Reach of Evidence-Based Practices to Support Student Attention and Behavior Through Technology — https://ies.ed.gov/funding/grantsearch/details.asp?ID=6036